CLINICAL TRIAL: NCT04001998
Title: A Two-Part, Open Label, Complete Crossover Study to Compare the Tablet and Capsule Formulations of BLD-2660, Including a Food Effect Assessment of the Tablet Formulation, and to Assess Dose Proportionality Following Single Oral Doses of BLD-2660 in Tablet Formulation
Brief Title: Healthy Volunteer Study Comparing Tablet and Capsule Formulations
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: On hold to determine chosen formulations
Sponsor: Blade Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B-2660-102
Record Dates: First submitted 2019-06-26; First posted 2019-06-28 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-09

CONDITIONS: Fibrosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet vs Capsule Formulation (Experimental): Single oral dose of BLD-2660 capsule or tablet formulation
  Interventions: Drug: BLD-2660
- Dose Proportionality (Experimental): Single oral dose of BLD-2660 tablet formulation
  Interventions: Drug: BLD-2660

INTERVENTIONS:
Drug: BLD-2660 — Randomized to active product

SUMMARY:
Single center, randomized, open label, two-part crossover study designed to evaluate the PK, food effect, dose proportionality, safety, and tolerability of BLD-2660 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Agree to no smoking or alcohol or illegal substance 48 hours prior to dosing
* Normal BMI (18 to ≤ 35 kg/m2)
* Have a negative urine drug screen/alcohol breath test on admission to clinic
* Agree to use highly effective, double barrier contraception (both male and female partners) during the study and for 90 days following completion of dosing
* Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine or serum pregnancy test on Day -1
* Be in general good health
* Clinical laboratory values within normal range

Exclusion Criteria:

* Recent wound, or presence of an ongoing non-healing skin wound
* Presence of any underlying physical or psychological medical condition that, in the opinion of the Investigator, would make it unlikely that the subject will complete the study per protocol
* History or presence of alcoholism or drug abuse within the 2 years prior to the first study drug administration, and unwillingness to be totally abstinent during the dosing period
* Blood donation or significant blood loss within 30 days prior to the first study drug administration
* Plasma donation within 7 days prior to the first study drug administration
* Administration of investigational product (IP) in another trial within 30 days prior to the first study drug administration, or five half-lives, whichever is longer
* Females who are pregnant or lactating
* Surgery within the past 3 months prior to the first study drug administration determined by the PI to be clinically relevant
* Failure to satisfy the PI of fitness to participate for any other reason
* Active infection or history of recurrent infections
* Active malignancy and history of malignancy in the past 2 years, with the exception of completely excised basal cell carcinoma or low grade cervical intraepithelial neoplasia
* Antibiotic treatment within 3 months
* Chronic medical condition
* Any acute illness within 30 days prior

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Area under the drug concentration-time curve from time zero to the last measurable concentration (AUC0-last) | Up to 40 days
  Measured by plasma concentration
AUC from time 0 to infinity (AUC0-inf) | Up to 40 days
  Measured by plasma concentration
Maximum observed drug concentration (Cmax) | Up to 40 days
  Measured by plasma concentration
Time of the maximum drug concentration (Tmax) | Up to 40 days
  Measured by plasma concentration
Apparent terminal half-life (t½) | Up to 40 days
  Measured by plasma concentration
Apparent terminal elimination rate constant (Kel) | Up to 40 days
  Measured by plasma concentration

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 40 days
  AEs will be assessed by determining the incidence, severity, and dose relationship of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Lemech, MD, Principal Investigator — Scientia Clinical Research
Locations (1):
- Scientia Clinical Research, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No